CLINICAL TRIAL: NCT03822143
Title: Fetus Anemia Diagnosis by Ultrasound Data Collection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0107-18
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Anemia in Fetus
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fetus anemia diagnosis (Experimental): Diagnosis of anemia in the fetus through use of ultrasound data collection
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Use of ultrasound device to diagnosis anemia in a fetus

SUMMARY:
The aim of this study is to diagnose anemia in fetuses through the use of ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 16th week to 41st week +6 days
* Singleton fetus

Exclusion Criteria:

* All others

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Anemia diagnosis in fetus | One week
  Data collection from use of ultrasound will be analyzed through a laboratory algorithm to determine whether a fetus has anemia

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No